CLINICAL TRIAL: NCT03651050
Title: Implementing a Digital Child Mental Health Screening, Literacy, and Management Tool in Faith-Based Settings
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: NYU Langone Health (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 18-00728
Record Dates: First submitted 2018-08-27; First posted 2018-08-29 (Actual); Last update posted 2021-12-09 (Actual); Status verified 2021-12

CONDITIONS: Mental Health
MeSH Terms: conditions — Psychological Well-Being | interventions — Community Health Workers

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- intervention FBOs receive the P-MHDT (Experimental)
  Interventions: Behavioral: Faith Based Outreach (FBO)
- control FBOs receive no P-MHDT (Experimental)
  Interventions: Behavioral: community-health-workers (CHW)

INTERVENTIONS:
Behavioral: Faith Based Outreach (FBO) — Faith base outreach groups will be trained in P-MHDT
  Arms: intervention FBOs receive the P-MHDT
Behavioral: community-health-workers (CHW) — COmmon health workers will be trained in P-MHDT
  Arms: control FBOs receive no P-MHDT

SUMMARY:
The proposed project is to develop a Pediatric-Mental Health Digital Toolkit (P-MHDT) Toolkit to support innovative child mental health preventive interventions in FBO settings. This project focuses on developing a P-MHDT and carrying out a pilot feasibility evaluation in real world settings. A group of Mental Health Professionals (MHPs)/ Community Healthcare Workers (CHWs) will be trained and the P-MHDT Toolkit intervention will be tested in 6 Faith Based Organizations (FBOs) in Uganda.

DETAILED DESCRIPTION:
The specific aims of this proposed study include:

Aim 1. To develop a P-MHDT (by employing qualitative focus-group interviews and user-centered design to enhance usability).

Aim 2. To train mental health professionals and community health workers (CHWs) for the P-MHDT approach of child mental health promotion in Uganda (including monitoring impacts of training on CHWs' program implementation competency).

Aim 3 (11-24 month). To estimate impacts of the P-MHDT on FBOs and families (i.e., caregivers' mental health literacy, practices, and children's mental health) when implemented in the real world FBO settings.

ELIGIBILITY:
Inclusion Criteria:

* Participants must be at least 18 years of age. Participating parents must be caregivers of age 1-7 years old children.
* Children are not the subjects of this study, and will not participate in research activities.

Exclusion Criteria:

* Evidence of psychopathology or cognitive impairment severe enough to preclude giving consent, or completing the survey instruments or the focus group of the study.
* Minors (age <18) will also be excluded.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 319 (Actual)
Dates: Start 2019-08-01 (Actual); Primary Completion 2020-08-30 (Actual); Study Completion 2021-08-01 (Actual)

PRIMARY OUTCOMES:
Aggression measured by parent report | 24 Months
Anxiety measured by parent report | 24 Months
Depression measured by parent report | 24 Months

CONTACTS AND LOCATIONS:
Overall Officials: Keng-Yen Huang, MD, Principal Investigator — NYU Langone Health
Locations (1):
- New York University Langone Health, New York, New York, United States